CLINICAL TRIAL: NCT07351357
Title: Multi-Centre Pragmatic Randomized Controlled Trial of Bowel Preparation Before Peritoneal Dialysis Catheter Insertion
Brief Title: Bisacodyl Oral for Lowering Dysfunction (of Tenckhoff Catheter)
Acronym: BOLD
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Chow Kai Ming, Dr, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CREC-2025-492
Record Dates: First submitted 2026-01-01; First posted 2026-01-20 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Renal Failure Chronic Requiring Dialysis; Peritoneal Dialysis
Keywords: peritoneal dialysis; Tenckhoff catheter; laxative; bowel preparation; catheter dysfunction
MeSH Terms: interventions — Bisacodyl

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bowel preparation (Active Comparator): oral bisacodyl
  Interventions: Drug: Bisacodyl 5 mg
- Usual care (No Intervention): usual care for catheter insertion

INTERVENTIONS:
Drug: Bisacodyl 5 mg — In the intervention arm, the protocol of prophylactic laxative is administration of oral enteric coated bisacodyl 5 mg at bedtime for two consecutive days prior to Tenckhoff catheter insertion. In the control arm, patients will receive usual care, and are allowed to continue their usual laxative, without extra prescription.
  Arms: Bowel preparation

SUMMARY:
Doctors need to insert catheter for patients who are going to have peritoneal dialysis. These peritoneal catheters can be obstructed or blocked afterward. The chance of not having smooth flow can be up to 12 and 31%. So far, constipation is one of the proposed reasons. Therefore, the study is aimed to investigate whether the preventive use of laxative before the surgery can help better improve the function of the catheter and hence better flow.

DETAILED DESCRIPTION:
This study compares the result of laxative bowel preparation versus usual care before the insertion of Tenckhoff catheters for peritoneal dialysis patients. The investigators design an open-label multi-centre randomized controlled study to evaluate the prophylactic use of laxative to reduce incidence of catheter flow dysfunction after peritoneal dialysis catheter insertion. The primary objective is to assess whether laxative prophylaxis can reduce the risk of catheter dysfunction that requires intervention. The investigators estimate that the study would need to enroll 199 peritoneal dialysis patients in each group for the study to have 80% power to detect a difference between 10% and 20% in the primary endpoint of catheter dysfunction requiring simple intervention.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 or older and need of peritoneal dialysis
* willingness to give written consent and comply with the study protocol

Exclusion Criteria:

* known contraindication to peritoneal dialysis
* ongoing diarrhoea or active inflammatory bowel disease
* participation in another interventional study within last 30 days of randomization
* history of a psychological illness or condition that would interfere with the patient's ability to understand the requirement of the study and/or comply with the dialysis procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 398 (Estimated)
Dates: Start 2026-01-12 (Estimated); Primary Completion 2027-08-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Catheter dysfunction | within 4 weeks of catheter insertion
  Primary outcome is the incidence of catheter dysfunction that requires simple and invasive manipulation by fluoroscopic or surgical procedure. Catheter dysfunction refers to drainage failure, as defined by the inability to drain peritoneal dialysate effluent reliably within 45 minutes. Simple intervention includes use of irrigation of catheter with saline, fibrinolytic agent such as urokinase and extra laxative use. Invasive manipulation of catheter includes repositioning or reinsertion, either by fluoroscopic method, open surgical or laparoscopic method.

SECONDARY OUTCOMES:
Catheter dysfunction and survival | 3 months after catheter insertion for early peritonitis
  The time to catheter dysfunction requiring invasive intervention
The incidence of early peritonitis (within 3 months of catheter insertion) | 3 months after catheter insertion
  Peritonitis
The peritoneal catheter survival | 3 months after catheter insertion
  catheter survival

CONTACTS AND LOCATIONS:
Locations (6):
- Hong Kong (6):
  - Princess Margaret Hospital, Kwai Chung, Kowloon
  - Caritas Medical Centre, Sham Shui Po, Kowloon
  - Prince of Wales Hospital, Shatin, NT
  - Tseung Kwan O Hospital, Tseung Kwan O, NT
  - Queen Elizabeth Hospital, Yau Ma Tei, NT
  - Prince of Wales Hospital, Shatin

IPD SHARING:
Plan to Share IPD: No
Confidentiality